CLINICAL TRIAL: NCT01916590
Title: Effectiveness of Continuous Femoral Nerve Block Versus Single Shot Femoral Nerve Block for Pain Control After Anterior Cruciate Ligament Reconstruction With Patellar Tendon Graft or Allograft
Brief Title: Effectiveness of Continuous Femoral Nerve Block Versus Single Shot Femoral Nerve Block for Pain Control
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of patients
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 11-0847
Record Dates: First submitted 2013-07-30; First posted 2013-08-05 (Estimated); Results first posted 2016-08-01 (Estimated); Last update posted 2016-08-01 (Estimated); Status verified 2016-06

CONDITIONS: Post-operative Pain
Keywords: Post-operative pain; Anterior Cruciate Ligament repair
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bupivacaine (Active Comparator): All patients who give consent will undergo ultrasound guided placement of a femoral catheter with injection of 30 cc of 0.5% bupivacaine (without epinephrine)through the catheter. After surgery before the patient is discharged home their femoral catheter will then be connected to the home pain pump filled with bupivacaine 0.25% solution (without epinephrine), and the infusion will be started at 6 ml/hr. gh the catheter.
  Interventions: Drug: Bupivicaine
- Placebo (Placebo Comparator): All patients who give consent will undergo ultrasound guided placement of a femoral catheter with injection of 30 cc of 0.5% bupivacaine (without epinephrine) through the catheter. After surgery before the patient is discharged home their femoral catheter will then be connected to the home pain pump filled with saline solution, and the infusion will be started at 6 ml/hr. gh the catheter.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Bupivicaine — After surgery before the patient is discharged home their femoral catheter will then be connected to the home pain pump filled with bupivacaine 0.25% solution (without epinephrine), and the infusion will be started at 6 ml/hr. gh the catheter.
  Arms: Bupivacaine
Drug: placebo
  Arms: Placebo

SUMMARY:
Both single shot femoral nerve block and continuous femoral nerve block with catheter have been shown to be effective for pain control after anterior cruciate ligament reconstruction (ACLR). Continuous femoral nerve block may be the more effective of the two in reducing pain scores and opioid consumption for the first 48 hours postoperatively.

DETAILED DESCRIPTION:
The number of ambulatory procedures has steadily increased over the last decade. Postoperative pain is the most common cause of delayed discharge and unexpected admission after ambulatory surgery. Knee surgery was identified as one of the procedures associated with the most pain at 24 hours, with a 45% or higher incidence of moderate or severe pain. Poor pain control can counteract many of the benefits of ambulatory surgery and can lead to the development of chronic pain.

Regional techniques have been shown to be effective after ACL reconstruction, allowing faster patient recovery with fewer side-effects than intravenous administration of opioids. Different regional techniques have been applied and studied after ACLR. Femoral nerve block for ACLR either as a single bolus or as a continuous infusion markedly decreases intravenous analgesic requirements and postoperative pain. To the Investigator's knowledge, no study has compared these two techniques after ACLR with patellar tendon graft or allograft.

ELIGIBILITY:
Inclusion Criteria:

1. American Society of Anesthesiologists score between 1-3
2. Scheduled to undergo Anterior Cruciate Ligament reconstruction with patellar tendon graft or allograft under general anesthesia

Exclusion Criteria:

1. Localized infection of the groin or generalized sepsis.
2. Hypersensitivity or known allergy to local anesthetics.
3. Preexisting nerve damage in surgical limb.
4. History of chronic pain with either (a) daily opioid requirement exceeding the equivalent of 50 mg morphine or (b) daily prescription of tricyclic antidepressants, gabapentin, pregabalin, or tramadol for pain.
5. Patients who elect to have knee surgery under spinal anesthesia or who cannot undergo general anesthetic.
6. Patients who decline to have a femoral nerve block with catheter.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2011-07; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Fiegel, M.D., Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Hospital, Aurora, Colorado, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: All patients who give consent will undergo ultrasound guided placement of a femoral catheter with injection of 30 cc of 0.5% bupivacaine (without epinephrine) through the catheter. After surgery before the patient is discharged home their femoral catheter will then be connected to the home pain pump filled with saline solution, and the infusion will be started at 6 ml/hr. gh the catheter.
  placebo
Period: Overall Study
Arm/Group | Bupivacaine | Placebo
Started | 4 | 3
Completed | 4 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bupivacaine | Placebo | Total
Number analyzed (Participants) | 4 | 3 | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 3 | 7
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 4 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: Pain Scores Will be Collected for 48 Hours After ACL Reconstruction
Description: Pain scores will be collected for 48 hours after ACL reconstruction with a patellar tendon graft or allograft and used to measure the effectiveness of the femoral catheter vs. single shot femoral nerve block
Time Frame: 48 hours after surgery
Population: Because of the lack of enrollment no data was collected
Arm/Group | Bupivacaine | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: Serious and Other (Not Including Serious) Adverse Events were not monitored/collected for the 7 enrolled participants.
Arm/Group | Bupivacaine | Placebo
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Serious and Other (Not Including Serious) Adverse Events were not monitored/collected for the 7 enrolled participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No